CLINICAL TRIAL: NCT03063268
Title: An Interactive Patient-Centered Consent for Research Using Medical Records
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Richard M. Fairbanks School of Public Health AT IUPUI (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB201602061 - N; R01HD086700 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Attitude to Computers; Attitude of Health Personnel; Researcher-Subject Relations; Trust; Communication Research
Keywords: Electronic Consent; Human Behavior; Bioethics; Research Ethics; Electronic Medical Records (EMR); Electronic Health Records (EHR); Informed Consent Form; Interactive Consent; Health Record Data

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trust-Enhanced Messaged with Interactive Features on E-Consent (Experimental): Messaging with trust-enhanced modification to the language that the research team has identified as beneficial additional knowledge to provide to participants. This messaging was reviewed by participants from Phase I and edited as suggested.
  Interventions: Behavioral: Trust-Enhanced Messaging on E-Consent; Behavioral: Interactive features on E-Consent; Behavioral: Standard E-Consent
- Interactive Features on E-Consent (Experimental): Interactive hyperlinks to open up to further information for key words that participants from Phase I and prototype design and testing have identified as gaps in subject knowledge and provision of information to subjects.
  Interventions: Behavioral: Interactive features on E-Consent; Behavioral: Standard E-Consent
- Standard E-Consent (Active Comparator): Standardized text currently used by the University of Florida (UF) IRB with no trust-enhanced messaging or interactive hyperlinks that provide further information for subjects.
  Interventions: Behavioral: Standard E-Consent

INTERVENTIONS:
Behavioral: Trust-Enhanced Messaging on E-Consent — Messaging with trust-enhanced modification to the language that the research team has identified as beneficial additional knowledge to provide to participants. This messaging was reviewed by participants from Phase I and edited as suggested.
  Other Names: Trust-Enhanced E-Consent
  Arms: Trust-Enhanced Messaged with Interactive Features on E-Consent
Behavioral: Interactive features on E-Consent — Interactive hyperlinks to open up to further information for key words that participants from Phase I and prototype design and testing have identified as gaps in subject knowledge and provision of information to subjects.
  Other Names: Interactive E-Consent
  Arms: Interactive Features on E-Consent; Trust-Enhanced Messaged with Interactive Features on E-Consent
Behavioral: Standard E-Consent — Standard consent currently used by the University of Florida (UF) IRB with no trust-enhanced messaging or interactive hyperlinks that provide further information for subjects.

SUMMARY:
The goal of this project is to develop and evaluate a novel, electronic informed consent application for research involving electronic health record (EHR) data. In response to NIH RFA-OD-15-002, this study addresses research using clinical records and data, including the issues of the appropriate content and duration of informed consent and patient preferences about research use of clinical information. This study will design an electronic consent application intended to improve patients' satisfaction with and understanding of consent for research using their EHR data. The electronic application will provide interactive functionality that creates a virtual, patient-centered discussion with patients about research that uses EHR data. Also, to correct potential misconceptions and increase informedness, the application will present trust-enhancing messages that highlight facts about research regulations, researcher training, and data protections. This study (Specific Aim 2 of the linked study protocol) will compare the effectiveness of the interactive, trust-enhanced consent application to an interactive consent and standard consent (no interactivity, no trust- enhancement) using a randomized trial of the three consents with 750 adults in a network of family medicine practices. Primary outcomes will be satisfaction with the consent decision and understanding of the consent content. This application will allow patients to learn more about clinical research and make informed choices about whether or not they want their health records and data to be used for research. This first phase of this project (IRB#:201500678) was innovative because it created a virtual, patient-centered discussion about research using EHR data. Moreover, this project produced a consent application that clinicians and researchers will use in this phase (Phase two) of the trial as an ethically sound and practical tool for consenting patients, in a clinical setting, for research involving EHRs. Overall, this study will improve understanding of how to best give patients information about research that uses their health records and data. With this understanding, this study will develop a new computer application that patients can use in their doctors' offices. This application will allow patients to learn more about clinical research and make informed choices about whether or not they want their health records and data to be used for research.

DETAILED DESCRIPTION:
This study (Specific Aim 2 of the linked study protocol) will compare the effectiveness of the interactive, trust-enhanced consent application to an interactive consent and standard consent (no interactivity, no trust- enhancement) using a randomized trial of the three consents with 750 adults in a network of family medicine practices. Primary outcomes will be satisfaction with the consent decision and understanding of the consent content.

Conceptually, the hypothesized effectiveness of this study's new consent application relies on two constructs, interactivity and trust. Many studies have identified the importance of trust in researchers when it comes to people's willingness to participate in research. Moreover, trust in the source of information is critical to participants' evaluations of risk information. And, risk information is an important element of the research consent process. Thus, highlighted relevant messages to participants at the outset of a research consent process. It is expected that these messages will not coerce participants nor will they dramatically alter participants' general trust in researchers. More importantly, empirically assessments of both of these expectations to ensure the application delivers an ethically appropriate consenting experience. However, it is expected that presenting key facts about research data protections, researcher training, and research regulations will increase the likelihood that participants will be willing to learn about research using medical records. In turn, this will increase participants' understanding and help them make a more informed decision. In the absence of these trust-related messages, it is expected that many participants will simply disengage from the details of the consent information and thus make a less informed decision about participating. Next, the investigators' use of interactivity is supported by research on the effectiveness of communications that interactively deliver detail, empower audiences, and allow a self - discovery process. Indeed, an interactive, person-to-person consent process is the standard approach in clinical trials. Therefore, in the new consent application, the interface will allow participants to interactively explore the details that are most important for their personal understanding of research using EHRs and most relevant to their personal information needs and satisfaction with the consent decision. Without this interactive information exploration, which is essentially dynamically tailored to their personal information needs, participants are more likely to be overwhelmed by the volume of information presented and unable to obtain the information they want most. Under these circumstances, participants' overall understanding of the consent information is likely to decrease, and they are likely to make less satisfactory decisions. There are two specific hypotheses: (1) compared to the standard consent, the interactive consent will lead to increased decisional satisfaction and understanding of the consent; and (2) compared to the interactive consent, the interactive, trust-enhanced consent will lead to increased decisional satisfaction and understanding of the consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a scheduled medical visit at a UF Family Medicine clinic
* Capacitated, english-speaking patients
* Ages 18 and over
* Patients who meets the above criteria and is willing to consent to participate in the trial.

Exclusion Criteria:

* Patients who do not complete the UF IRB approved informed consent form
* Patients under the age of 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Baseline Satisfaction with consent decision | Immediate at baseline
  Satisfaction With Decisions scale (Holmes-Rovner et al. 1996); 6-items, 5-point Likert scale (strongly disagree-strongly agree)
Change from Baseline Satisfaction with consent decision | 1-week follow-up from Baseline
  Satisfaction With Decisions scale (Holmes-Rovner et al. 1996); 6-items, 5-point Likert scale (strongly disagree-strongly agree)
Baseline Understanding of consent content | Immediate at Baseline
  Modified version of the Quality of Informed Consent scale, Part B (Joffe et al. 2001); 14-items, 5-point Likert scale (I didn't understand this at all - I understood this very well)*
Change from Baseline Understanding of consent content | 1-week follow-up from Baseline
  Modified version of the Quality of Informed Consent scale, Part B (Joffe et al. 2001); 14-items, 5-point Likert scale (I didn't understand this at all - I understood this very well)*
Change from Baseline Understanding of consent content | 6-month follow-up from Baseline
  Modified version of the Quality of Informed Consent scale, Part B (Joffe et al. 2001); 14-items, 5-point Likert scale (I didn't understand this at all - I understood this very well)*

SECONDARY OUTCOMES:
Baseline Perceived Voluntariness | Immediate at Baseline
  Decision Making Control instrument to assess voluntary consent (Miller et. al.,2011); 9-items, 5-point Likert Scale (Strongly disagree-Strongly Agree)
Change from Baseline Perceived Voluntariness | 1-week follow-up from Baseline
  Decision Making Control instrument to assess voluntary consent (Miller et. al.,2011); 9-items, 5-point Likert Scale (Strongly disagree-Strongly Agree)
Baseline Trust in medical researchers | Prior to consent
  Trust In Medical Researchers Scale (Mainous et al. 2006); 12 items, 5-point Likert scale (strongly disagree-strongly agree); Aggregate scores range from 0-48 Sub-analysis of the two Trust in Medical Researchers subscales (or TIMRS)- Participant Deception; Researcher Honesty.
Change from Baseline Trust in medical researchers | Immediate at Baseline
  Trust In Medical Researchers Scale (Mainous et al. 2006); 12 items, 5-point Likert scale (strongly disagree-strongly agree); Aggregate scores range from 0-48 Sub-analysis of the two Trust in Medical Researchers subscales (or TIMRS)- Participant Deception; Researcher Honesty.
Change from Baseline Trust in medical researchers | 1-week follow-up from Baseline
  Trust In Medical Researchers Scale (Mainous et al. 2006); 12 items, 5-point Likert scale (strongly disagree-strongly agree); Aggregate scores range from 0-48 Sub-analysis of the two Trust in Medical Researchers subscales (or TIMRS)- Participant Deception; Researcher Honesty.
Change from Baseline Trust in medical researchers | 6-month follow-up from Baseline
  Trust In Medical Researchers Scale (Mainous et al. 2006); 12 items, 5-point Likert scale (strongly disagree-strongly agree); Aggregate scores range from 0-48 Sub-analysis of the two Trust in Medical Researchers subscales (or TIMRS)- Participant Deception; Researcher Honesty.
Baseline Willingness to participate in research (i.e., allow EHR to be used in research); | Immediate at Baseline
  Consent for past and future EHR data to be shared with researchers for IRB-approved studies (yes/no); Consent for EHR to be linked with biospecimen data and released to researchers (yes/no)
Change from Baseline Willingness to participate in research (i.e., allow EHR to be used in research); | 1-week follow-up from Baseline
  Consent for past and future EHR data to be shared with researchers for IRB-approved studies (yes/no); Consent for EHR to be linked with biospecimen data and released to researchers (yes/no)
Change from Baseline Willingness to participate in research (i.e., allow EHR to be used in research); | 6-month follow-up from Baseline
  Consent for past and future EHR data to be shared with researchers for IRB-approved studies (yes/no); Consent for EHR to be linked with biospecimen data and released to researchers (yes/no)
Engagement with consent information | Immediate at Baseline (only)
  Time spent using consent application and click activity; Focused immersion in information (Agarwal & Karahanna 2000); 5 items, 5-point Likert scale (strongly disagree-strongly agree)
Baseline Numeracy Abilities | Immediate at Baseline
  Level of comfort, understanding, and preferences regarding commonly used mathematical skills (percentages, ratios, and probability)
Change from Baseline Numeracy Abilities | 1-week follow-up from Baseline
  Level of comfort, understanding, and preferences regarding commonly used mathematical skills (percentages, ratios, and probability)
Change from Baseline Numeracy Abilities | 6-month follow-up from Baseline
  Level of comfort, understanding, and preferences regarding commonly used mathematical skills (percentages, ratios, and probability)
Baseline Possibility of using a Computer Application | Immediate at Baseline
  Ease of use, comfort with, and improvements associated with Computer application use
Change from Baseline Possibility of using a Computer Application | 1-week follow-up from Baseline
  Ease of use, comfort with, and improvements associated with Computer application use
Change from Baseline Possibility of using a Computer Application | 6-month follow-up from Baseline
  Ease of use, comfort with, and improvements associated with Computer application use
Baseline Using new Computer Applications | Immediate at Baseline
  Experiences with computer applications that the participant has never used before
Change from Baseline Using new Computer Applications | 1-week follow-up from Baseline
  Experiences with computer applications that the participant has never used before
Change from Baseline Using new Computer Applications | 6-month follow-up from Baseline
  Experiences with computer applications that the participant has never used before
Baseline Dissemination & Access of Personal Health Records and Health Information | Immediate at Baseline
  Sharing of personal health record information with trusted scientists, healthcare providers, and past experiences of accessing personal health records
Change from Baseline Dissemination & Access of Personal Health Records and Health Information | 1-week follow-up from Baseline
  Sharing of personal health record information with trusted scientists, healthcare providers, and past experiences of accessing personal health records
Change from Baseline Dissemination & Access of Personal Health Records and Health Information | 6-month follow-up from Baseline
  Sharing of personal health record information with trusted scientists, healthcare providers, and past experiences of accessing personal health records

CONTACTS AND LOCATIONS:
Overall Officials: Ray E Moseley, Ph.D, Principal Investigator — University of Florida- College of Medicine- Department of Community Health & Family Medicine; Christopher A Harle, Ph.D, Principal Investigator — Indiana University- Purdue University Indianapolis- Richard M. Fairbanks School of Public Health; Arch G Mainous, Ph.D, Principal Investigator — University of Florida- Department of Health Services Research, Management and Policy
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harle CA, Golembiewski EH, Rahmanian KP, Brumback B, Krieger JL, Goodman KW, Mainous AG, Moseley RE. Does an interactive trust-enhanced electronic consent improve patient experiences when asked to share their health records for research? A randomized trial. J Am Med Inform Assoc. 2019 Jul 1;26(7):620-629. doi: 10.1093/jamia/ocz015. PMID 30938751